CLINICAL TRIAL: NCT04088227
Title: Effect of Platelet Rich Plasma Injections on Inflammatory and Chondrodegenerative Biomarkers in Patients With Acute Anterior Cruciate Ligament Tears
Brief Title: Effects of Platelet Rich Plasma Injections on Biomarkers After Anterior Cruciate Ligament Tears
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACL-PRP Study
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The control group will have a joint aspiration performed at an initial visit (within the first 10 days after injury), and at the time of surgery (within 4 weeks of injury).
  Interventions: Other: Control Group
- Experimental Group (Experimental): The experimental group will have a joint aspiration performed at an initial visit (within the first 10 days after injury) and receive an injection of leukocyte poor platelet rich plasma injection in their knee. At a second visit 5-12 days after the initial visit, the patient will receive a joint aspiration and platelet rich plasma injection. A final joint aspiration will be performed at the time of surgery (within 4 weeks of injury).
  Interventions: Drug: Experimental Group

INTERVENTIONS:
Drug: Experimental Group — Patients will receive platelet rich plasma injection two times prior to surgery.
  Other Names: Platelet Rich Plasma
  Arms: Experimental Group
Other: Control Group — Patients will have their knee aspirated at their initial physician visit and at the time of surgery.
  Other Names: Aspiration Only
  Arms: Control Group

SUMMARY:
A potential long-term consequence of anterior cruciate ligament injuries is the development of post-traumatic osteoarthritis in the years following injury. There are no curative treatments for osteoarthritis, increasing the importance of minimizing the occurrence of post-traumatic osteoarthritis following anterior cruciate ligament injuries. Current literature has begun to indicate that biochemical changes in the knee joint cartilage, such as chondrocyte death, following injury can contribute to the development of post-traumatic osteoarthritis.

The main objective of this study is to determine if an early intervention of joint aspiration and platelet rich plasma injection will positively affect the biomarkers representative of chondral degeneration in patients with anterior cruciate ligament injuries. We hypothesize that the intervention will reduce the volume of inflammatory and chondrodegenerative biomarkers following anterior cruciate ligament injury.

DETAILED DESCRIPTION:
A non-surgical treatment option for the management of osteoarthritis include injectables such as corticosteroids and platelet rich plasma. These injectables work by positively affecting cartilage cells, also known as chondrocytes, and the cells of the joint lining tissue, also known as synoviocytes. Platelet rich plasma is an autologous derived blood product, i.e. a joint injectable made from the patient's own blood at the time and location of injection with simple blood centrifugation. Studies in the bench-top laboratory setting have provided in-vitro evidence that platelet rich plasma decreases synoviocyte production of metallometal proteases, an inflammatory protein with negative effects on cartilage and decreases the effects of inflammatory proteins.

ELIGIBILITY:
Inclusion Criteria:

* No history of previous traumatic ipsilateral knee injury
* Bone bruise visualized on MRI
* No clinical evidence of posterior cruciate ligament injury with no more than grade 1 medial or lateral collateral ligament injury

Exclusion Criteria:

* Patients without a palpable knee effusion
* An injury occurring more than 10 days before enrollment
* Previous ipsilateral knee surgery
* Intra-articular cortisone or platelet rich plasma injection into either knee within 3 months of injury
* Participation in another clinical drug trial within the 4 weeks before injury
* A history of any inflammatory disease or immune-comprised

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Anz, MD, Principal Investigator — Andrews Institute for Orthopaedics & Sports Medicine
Locations (1):
- Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anz AW, Branch EA, Jordan SE, Ostrander RV 3rd, Kindle BJ, Presley JC, Hackel JG, Maggi E, Plummer HA. Preoperative Platelet-Rich Plasma Injections Decrease Inflammatory and Chondrodegenerative Biomarkers in Patients With Acute Anterior Cruciate Ligament Tears: A Pilot Randomized Controlled Trial. Orthop J Sports Med. 2025 Mar 3;13(3):23259671241312754. doi: 10.1177/23259671241312754. eCollection 2025 Mar. PMID 40052182

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Surgery postponed >5weeks | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (8) | 20 (6.7) | 20 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] | 87.6 (26.7) | 68.5 (12.8) | 80.8 (21.56)
Height [Mean (Standard Deviation); unit: cm] | 173 (11.5) | 174.6 (8.3) | 174.6 (11.63)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (6.8) | 22.5 (4) | 26.2 (6.48)
Time to Surgery (days) [Mean (Standard Deviation); unit: days] | 16.9 (6.8) | 27 (13.1) | 20.74 (9.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in Synovial Interleukin (IL) -1 Receptor Antagonist Concentration
Description: The presence of the Synovial Interleukin (IL) -1 Receptor Antagonist biomarker in the synovial fluid will be assessed.
Time Frame: Timepoint 1: initial visit (within 10 days of injury) Timepoint 2: at the time of surgery (within 4 weeks of injury)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 12 | 12
pg/ml
  IL-1ß Timepoint 1 | 13.8 (4.1) | 16 (4.9)
  IL-1ß Timepoint 2 | 9.9 (4.9) | 7.5 (4.5)
  IL-10 Timepoint 1 | 53.1 (16.4) | 64.3 (21.4)
  IL-10 Timepoint 2 | 36.1 (20.3) | 31.7 (19.2)
  IL-6 Timepoint 1 | 7668.6 (4092.9) | 8650.8 (3983.9)
  IL-6 Timepoint 2 | 3940.2 (3809.2) | 2196.2 (2994.2)
  GM- CSF Timepoint 1 | 20.6 (7.1) | 25.3 (9.1)
  GM- CSF Timepoint 2 | 16 (10.1) | 12.4 (9.5)
  IL-5 Timepoint 1 | 30.6 (16.7) | 48.8 (23.9)
  IL-5 Timepoint 2 | 27.9 (23.3) | 24.7 (19.7)
  IFN-γ Timepoint 1 | 2.5 (1.1) | 4.0 (1.7)
  IFN-γ Timepoint 2 | 2.6 (1.5) | 1.7 (1.3)
  TNF-⍺ Timepoint 1 | 11.2 (7.0) | 21.6 (9.5)
  TNF-⍺ Timepoint 2 | 10.4 (9.1) | 10.9 (7.9)
  IL-2 Timepoint 1 | 29.2 (24.9) | 54.6 (34.3)
  IL-2 Timepoint 2 | 32.7 (32.5) | 28.6 (25.9)
  IL-4 Timepoint 1 | 278.2 (144.4) | 398.5 (189.4)
  IL-4 Timepoint 2 | 234.5 (161.6) | 200.2 (167.7)
  IL-8 Timepoint 1 | 315.1 (80.3) | 1295.2 (1075.9)
  IL-8 Timepoint 2 | 124.8 (49.7) | 222.6 (113.4)

ADVERSE EVENTS:
Time Frame: One year per standard of care after ACL injury.
Arm/Group | Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04088227/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04088227/ICF_001.pdf